CLINICAL TRIAL: NCT03795961
Title: Evaluation of The Neuromedulatory Effect of Transcranial Direct Current Electrical Stimulation (tDCS) in Carpal Tunnel Syndrome (CTS): A Double Blinded Randomized Clinical Trial
Brief Title: Neuromedulatory Effect of Transcranial Direct Current Electrical Stimulation in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Gehad Swilam Abdelmonem Swilam, Assistant Lecturer, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSMGAEAM
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: the study subject will be allocated into two group ; active and sham group
Who Masked: Participant, Outcomes Assessor
Masking Description: To make sure that no bias should enter the assessment of the results, neither the patient nor the clinicians will be aware whether active tDCS will be applicated to a particular case. To ensure this result, two symbols (Square and Triangle) will be applicated to the physiotherapy sheet and only the physiotherapist knew the key for each symbol. The triangle may represent the cases of CTS for active tDCS and the square may represent the sham group or vice versa. At the end of the study the two groups will be revealed in order to analyze the results according to proper statistical measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS group (Experimental): This group will include 42 patients with CTS Intervention (active transcranial direct current electrical stimulation) Stimulation site (M1) Stimulation mode (anodal) Duration of session (20 minutes) Stimulation intensity (2 mA) Number of sessions (5 sessions) Intervals (every another day)
  Interventions: Device: transcranial direct current electrical stimulation
- Sham tDCS group (Sham Comparator): This group will include 42 patients with CTS Intervention (sham or inactive transcranial direct current electrical stimulation) Stimulation site (M1) Stimulation mode (anodal) Duration of session (20 minutes) Stimulation intensity (2 mA) Number of sessions (5 sessions) Intervals (every another day)
  Interventions: Device: transcranial direct current electrical stimulation

INTERVENTIONS:
Device: transcranial direct current electrical stimulation — anodal tDCS of M1 for 20 minutes, at 2 mA for 5 sessions (day after day)

SUMMARY:
This is a double blinded randomized clinical trial to study the neuromodulatory effect of tDCS in patients with CTS, the study subject will be randomly into two groups; active and sham group , the active group will receive five sessions of active TDCS over the M1 while the Sham group will receive sham tDCS in which the device will be turned off after 30 seconds. The patient will be assessed by VAS score, Boston carpal tunnel questionnaire , central sensetization inventory , pressure pain threshold, sensory and pain threshold for electerical stimulation before , after the end of the sessions and 4 weeks later.

DETAILED DESCRIPTION:
The study will be carried out on patients attending the Physical Medicine, Rheumatology and Rehabilitation outpatient clinic in Suez Canal University Hospital, Ismailia, EGYPT and diagnosed with CTS according to clinical examination and to the American Association of Neuromuscular and Electrodiagnostic Medicine (AANEM) practice recommendations for CTS.

Study subjects will be divided into two groups:

Group (1): (active group) will include 42 patients with CTS and will receive anodal tDCS of M1 for 20 minutes, at 2 mA for 5 sessions and less than 72 hrs. may be allowed between experimental sessions for each participant to avoid any interference.

Group (2): (sham group) will include 42 patients with CTS and will receive sham tDCS M1 (the set will be turned off after 30 seconds) for 20 minutes, at 2 mA for 5 sessions.

The study sample will be collected from all patients with CTS attending to the Physical medicine, Rheumatology and Rehabilitation outpatient clinic in Suez Canal University Hospital fulfilling the eligibility criteria, will be eligible to join the study (either referred for electrophysiological study or presented to the clinic for primary assessment). To make sure that no bias should enter the assessment of the results, neither the patient nor the clinicians will be aware whether active tDCS will be applicated to a particular case. To ensure this result, two symbols (Square and Triangle) will be applicated to the physiotherapy sheet and only the physiotherapist knew the key for each symbol. The triangle may represent the cases of CTS for active tDCS and the square may represent the sham group or vice versa. At the end of the study the two groups will be revealed in order to analyze the results according to proper statistical measures.

ELIGIBILITY:
Inclusion Criteria:

Patient diagnosed as CTS by history, clinical examination and NCS for more than 3 months.

Both genders. Adult of aged 18 years and above. Able to understand the informed consent.

Exclusion Criteria:

Patients with diabetes mellitus, collagen disorders, thyroid disease, peripheral neuropathy, traumatic nerve injury, cervical radiculopathy, fibromyalgia.

Pregnancy. Malignant. Patients with any clinically significant or unstable medical or psychiatric disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-12-16 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | before sessions (baseline assessment)
  Visual analogue scale is a measurement instrument that measure the pain across a continuum of values. Visual analogue scale is measured in millimeters and ranged from minimum (0 millimeter) to maximum (100 millimeters), where, score 0 indicates no pain and 100 indicates worst pain ever.
Visual analogue scale (VAS) | immediately after the ending of sessions
  Visual analogue scale is a measurement instrument that measure the pain across a continuum of values. Visual analogue scale is measured in millimeters and ranged from minimum (0 millimeter) to maximum (100 millimeters), where, score 0 indicates no pain and 100 indicates worst pain ever.
Visual analogue scale (VAS) | four weeks after the ending of sessions
  Visual analogue scale is a measurement instrument that measure the pain across a continuum of values. Visual analogue scale is measured in millimeters and ranged from minimum (0 millimeter) to maximum (100 millimeters), where, score 0 indicates no pain and 100 indicates worst pain ever.
Sensory threshold and pain threshold for electrical stimulation | before sessions (baseline assessment)
  Electrical stimulation will be applied by a pen electrode (model: 2762CC; Chattanooga) to the median nerve (pulse duration - 200 microseconds) at wrist level. Current supply start at 0 milli-ampere and will be increased in steps of 0.1 milli-ampere, until the participant report sensation and pain. The intensity of current (in milli-ampere) at which perception of the electrical stimulus first reported will be taken as sensory threshold; the intensity of current (in milli-ampere) at which participants first reported pain will be taken as pain threshold. These measurements will be averaged for analysis. Both sides will be assessed and compared. The lower the intensity of current (in milli-ampere) perceived, the worse the threshold, while the higher the intensity of current (in milli-ampere) perceived, the better the threshold.
Sensory threshold and pain threshold for electrical stimulation | immediately after the ending of sessions
  Electrical stimulation will be applied by a pen electrode (model: 2762CC; Chattanooga) to the median nerve (pulse duration - 200 microseconds) at wrist level. Current supply start at 0 milli-ampere and will be increased in steps of 0.1 milli-ampere, until the participant report sensation and pain. The intensity of current (in milli-ampere) at which perception of the electrical stimulus first reported will be taken as sensory threshold; the intensity of current (in milli-ampere) at which participants first reported pain will be taken as pain threshold. These measurements will be averaged for analysis. Both sides will be assessed and compared. The lower the intensity of current (in milli-ampere) perceived, the worse the threshold, while the higher the intensity of current (in milli-ampere) perceived, the better the threshold.
Sensory threshold and pain threshold for electrical stimulation | four weeks after the ending of sessions
  Electrical stimulation will be applied by a pen electrode (model: 2762CC; Chattanooga) to the median nerve (pulse duration - 200 microseconds) at wrist level. Current supply start at 0 milli-ampere and will be increased in steps of 0.1 milli-ampere, until the participant report sensation and pain. The intensity of current (in milli-ampere) at which perception of the electrical stimulus first reported will be taken as sensory threshold; the intensity of current (in milli-ampere) at which participants first reported pain will be taken as pain threshold. These measurements will be averaged for analysis. Both sides will be assessed and compared. The lower the intensity of current (in milli-ampere) perceived, the worse the threshold, while the higher the intensity of current (in milli-ampere) perceived, the better the threshold.
Pressure pain threshold assessment | before sessions (baseline assessment)
  Pressure will be induced using a pressure algometer (PainTest™ FPN 100 Algometer (Wagner Instruments, Greenwich, USA)) with a flat circular metal probe dressed in a rubber cover with a surface area of 1 cm2 applied to median, ulnar, radial, and c5-6 zygoapophyseal joint, The algometer will be mounted vertically and the pressure will be increased. Patients are asked to notify the investigator when they start to feel pain (pain threshold). For each measurement the algometer will be calibrated to enable force to be applied at a controlled and steady rate, the mean of three trials (intra-examiner reliability) will be calculated and used for main analysis. A 30 seconds resting period will be allowed between each measure. Both sides will be assessed and compared. Abnormal pressure pain threshold is at least 2 kg/cm2 different than that of the opposite site. The lower the value perceived, the worse the threshold, while the higher the value perceived, the better the threshold.
Pressure pain threshold assessment | immediately after the ending of sessions
  Pressure will be induced using a pressure algometer (PainTest™ FPN 100 Algometer (Wagner Instruments, Greenwich, USA)) with a flat circular metal probe dressed in a rubber cover with a surface area of 1 cm2 applied to median, ulnar, radial, and c5-6 zygoapophyseal joint, The algometer will be mounted vertically and the pressure will be increased. Patients are asked to notify the investigator when they start to feel pain (pain threshold). For each measurement the algometer will be calibrated to enable force to be applied at a controlled and steady rate, the mean of three trials (intra-examiner reliability) will be calculated and used for main analysis. A 30 seconds resting period will be allowed between each measure. Both sides will be assessed and compared. Abnormal pressure pain threshold is at least 2 kg/cm2 different than that of the opposite site. The lower the value perceived, the worse the threshold, while the higher the value perceived, the better the threshold.
Pressure pain threshold assessment | four weeks after the ending of sessions
  Pressure will be induced using a pressure algometer (PainTest™ FPN 100 Algometer (Wagner Instruments, Greenwich, USA)) with a flat circular metal probe dressed in a rubber cover with a surface area of 1 cm2 applied to median, ulnar, radial, and c5-6 zygoapophyseal joint, The algometer will be mounted vertically and the pressure will be increased. Patients are asked to notify the investigator when they start to feel pain (pain threshold). For each measurement the algometer will be calibrated to enable force to be applied at a controlled and steady rate, the mean of three trials (intra-examiner reliability) will be calculated and used for main analysis. A 30 seconds resting period will be allowed between each measure. Both sides will be assessed and compared. Abnormal pressure pain threshold is at least 2 kg/cm2 different than that of the opposite site. The lower the value perceived, the worse the threshold, while the higher the value perceived, the better the threshold.

SECONDARY OUTCOMES:
Boston carpal tunnel syndrome questionnaire | before sessions (baseline assessment)
  Boston carpal tunnel syndrome questionnaire is a disease-specific measure of self-reported symptom severity and functional status. It is frequently used in the reporting of outcomes from trials into interventions for carpal tunnel syndrome. Boston carpal tunnel syndrome questionnaire contains two sub-scales: symptom severity scale (11 items) and functional status scale (8 items). Scoring instructions: add the numbers corresponding to all answers and divide by the number of questions answered. Composite score (round to nearest 1/100th). The scores of symptom severity scale is ranged from 1-5, where, score 1 indicates no pain and score 5 indicates very severe pain. The scores of functional status scale is ranged from 1-5, where, score 1 indicates no difficulty and score 5 indicates cannot do at all due to hand or wrist.
Boston carpal tunnel syndrome questionnaire | immediately after the ending of sessions
  Boston carpal tunnel syndrome questionnaire is a disease-specific measure of self-reported symptom severity and functional status. It is frequently used in the reporting of outcomes from trials into interventions for carpal tunnel syndrome. Boston carpal tunnel syndrome questionnaire contains two sub-scales: symptom severity scale (11 items) and functional status scale (8 items). Scoring instructions: add the numbers corresponding to all answers and divide by the number of questions answered. Composite score (round to nearest 1/100th). The scores of symptom severity scale is ranged from 1-5, where, score 1 indicates no pain and score 5 indicates very severe pain. The scores of functional status scale is ranged from 1-5, where, score 1 indicates no difficulty and score 5 indicates cannot do at all due to hand or wrist.
Boston carpal tunnel syndrome questionnaire | four weeks after the ending of sessions
  Boston carpal tunnel syndrome questionnaire is a disease-specific measure of self-reported symptom severity and functional status. It is frequently used in the reporting of outcomes from trials into interventions for carpal tunnel syndrome. Boston carpal tunnel syndrome questionnaire contains two sub-scales: symptom severity scale (11 items) and functional status scale (8 items). Scoring instructions: add the numbers corresponding to all answers and divide by the number of questions answered. Composite score (round to nearest 1/100th). The scores of symptom severity scale is ranged from 1-5, where, score 1 indicates no pain and score 5 indicates very severe pain. The scores of functional status scale is ranged from 1-5, where, score 1 indicates no difficulty and score 5 indicates cannot do at all due to hand or wrist.
Central sensitization inventory | before sessions (baseline assessment)
  Central sensitization inventory is a screening instrument for clinicians to help identify patients with central sensitivity syndrome. Central sensitization inventory consists of two parts. Part A, one is asked how often he/she experiences each symptom ("never, rarely, sometimes, often, or always"). Individual items are scored from "0" (never) to "4" (always), resulting in a total score range for all 25 items from "0" to "100." A score of 40 or higher indicates the presence of central sensitivity syndrome. Part B asked if one has been previously diagnosed with seven common central sensitivity syndrome diagnoses (tension headaches/migraines, fibromyalgia, irritable bowel syndrome, restless leg syndrome, temporomandibular joint disorder, chronic fatigue syndrome, and multiple chemical sensitivities) and three central sensitization-related diagnoses (depression, anxiety/panic attacks, and neck injury). Central sensitization inventory B is for information only and is not scored.
Central sensitization inventory (CSI) | immediately after the ending of sessions
  Central sensitization inventory is a screening instrument for clinicians to help identify patients with central sensitivity syndrome. Central sensitization inventory consists of two parts. Part A, one is asked how often he/she experiences each symptom ("never, rarely, sometimes, often, or always"). Individual items are scored from "0" (never) to "4" (always), resulting in a total score range for all 25 items from "0" to "100." A score of 40 or higher indicates the presence of central sensitivity syndrome. Part B asked if one has been previously diagnosed with seven common central sensitivity syndrome diagnoses (tension headaches/migraines, fibromyalgia, irritable bowel syndrome, restless leg syndrome, temporomandibular joint disorder, chronic fatigue syndrome, and multiple chemical sensitivities) and three central sensitization-related diagnoses (depression, anxiety/panic attacks, and neck injury). Central sensitization inventory B is for information only and is not scored.
Central sensitization inventory (CSI) | four weeks after the ending of sessions
  Central sensitization inventory is a screening instrument for clinicians to help identify patients with central sensitivity syndrome. Central sensitization inventory consists of two parts. Part A, one is asked how often he/she experiences each symptom ("never, rarely, sometimes, often, or always"). Individual items are scored from "0" (never) to "4" (always), resulting in a total score range for all 25 items from "0" to "100." A score of 40 or higher indicates the presence of central sensitivity syndrome. Part B asked if one has been previously diagnosed with seven common central sensitivity syndrome diagnoses (tension headaches/migraines, fibromyalgia, irritable bowel syndrome, restless leg syndrome, temporomandibular joint disorder, chronic fatigue syndrome, and multiple chemical sensitivities) and three central sensitization-related diagnoses (depression, anxiety/panic attacks, and neck injury). Central sensitization inventory B is for information only and is not scored.

CONTACTS AND LOCATIONS:
Overall Officials: Mona S Ghaly, MD, Study Director — Suez Canal University
Locations (1):
- Suez Canal University Hospital, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD are not to be shared with other researchers